CLINICAL TRIAL: NCT02305017
Title: Effect of Paracetamol on Opicapone Pharmacokinetics in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BIA-91067-125
Record Dates: First submitted 2014-11-28; First posted 2014-12-02 (Estimated); Results first posted 2015-11-18 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-10

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — opicapone; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Period 1 OPC + Paracetamol; Period 2 OPC (Experimental): Period 1 BIA 9-1067 (Opicapone, OPC) + Paracetamol; Period 2 BIA 9-1067 (Opicapone, OPC)
  Interventions: Drug: BIA 9-1067; Drug: Paracetamol
- Period 1 OPC; Period 2 OPC+ Paracetamol (Experimental): Period 1 BIA 9-1067 (Opicapone, OPC) Period 2 BIA 9-1067 (Opicapone, OPC) + Paracetamol;
  Interventions: Drug: BIA 9-1067; Drug: Paracetamol

INTERVENTIONS:
Drug: BIA 9-1067 — BIA 9-1067 50 mg
  Other Names: OPC, Opicapone
Drug: Paracetamol — Paracetamol 1g
  Other Names: acetaminophen

SUMMARY:
Single-centre, open-label, randomised, two-way cross-over study consisting of 2 periods separated by a washout period of 14 days or more.

DETAILED DESCRIPTION:
Single-centre, open-label, randomised, two-way cross-over study consisting of 2 periods separated by a washout period of 14 days or more. In one period, subjects received three single-doses of 1 g paracetamol separated by 6 hours and 1.5 hours after the last paracetamol dose a single-dose of 50 mg OPC was administered.In the other period, a single-dose of 50 mg OPC was administered alone.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are able and willing to give written informed consent.
* Male or female subjects aged between 18 and 45 years, inclusive.
* Subjects of body mass index (BMI) between 19.0 and 30.0 kg/m2, inclusive.
* Subjects who are healthy as determined by pre-study medical history, physical examination, vital signs, complete neurological examination and 12-lead ECG.
* Subjects who have negative tests for HBsAg, anti-HCVAb and HIV-1 and HIV-2 Ab at screening.
* Subjects who have clinical laboratory test results clinically acceptable at screening and admission to each treatment period.
* Subjects who have a negative screen for alcohol and drugs of abuse at screening and admission to each treatment period.
* Subjects who are non-smokers or ex-smokers for at least 3 months.
* (If female) She is not of childbearing potential by reason of surgery or, if of childbearing potential, she uses an effective non-hormonal method of contraception (intrauterine device or intrauterine system; condom or occlusive cap [diaphragm or cervical or vault caps] with spermicidal foam or gel or film or cream or suppository; true abstinence; or vasectomized male partner, provided that he is the sole partner of that subject) for all the duration of the study.
* (If female) She has a negative serum pregnancy test at screening and a negative urine pregnancy test on Day -1 of each treatment period.

Exclusion Criteria:

* Subjects who have a clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine, connective tissue diseases or disorders.
* Subjects who have a clinically relevant surgical history.
* Subjects who have any clinically relevant abnormality in the coagulation tests.
* Subjects who have any clinically relevant abnormality in the liver function tests (a case-by-case decision for any abnormality must be discussed with the Sponsor before inclusion).
* Subjects who have a history of relevant atopy or drug hypersensitivity, particularly to paracetamol or any COMT inhibitor.
* Subjects who have a history of alcoholism or drug abuse.
* Subjects who consume more than 14 units of alcohol a week.
* Subjects who have a significant infection or known inflammatory process at screening or admission to each treatment period.
* Subjects who have acute gastrointestinal symptoms (e.g., nausea, vomiting, diarrhoea, heartburn) at the time of screening or admission to each treatment period.
* Subjects who have received paracetamol within 2 weeks of admission to the first period.
* Subjects who have used any other medicines within 2 weeks of admission to first period that may affect the safety or other study assessments, in the investigator's opinion.
* Subjects who have previously received OPC.
* Subjects who have used any investigational drug or participated in any clinical trial within 90 days prior to screening.
* Subjects who have participated in more than 2 clinical trials within the 12 months prior to screening.
* Subjects who have donated or received any blood or blood products within the 3 months prior to screening.
* Subjects who are vegetarians, vegans or have medical dietary restrictions.
* Subjects who cannot communicate reliably with the investigator.
* Subjects who are unlikely to co-operate with the requirements of the study.
* Subjects who are unwilling or unable to give written informed consent.
* (If female) She is pregnant or breast-feeding.
* (If female) She is of childbearing potential and she does not use an approved effective contraceptive method or she uses oral contraceptives.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2014-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Period 1 OPC + Paracetamol; Period 2 OPC | Period 1 OPC; Period 2 OPC+ Paracetamol
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Period 1 OPC + Paracetamol; Period 2 OPC | Period 1 OPC; Period 2 OPC+ Paracetamol | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 14 | 28
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Plasma Concentration
Description: Cmax - Maximum plasma concentration of opicapone on Day 12 following an oral single-dose of 50 mg OPC administered alone or 1.5 h after last 1 g Paracetamol administration
Time Frame: before and ½, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hour post-OPC dose
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Opicapone Alone: Opicapone, OPC, BIA 9-1079 alone
- Opicapone Plus Paracetamol: Opicapone, OPC, BIA 9-1079 Paracetamol acetominophen
Arm/Group | Opicapone Alone | Opicapone Plus Paracetamol
Number analyzed (Participants) | 28 | 28
ng/mL | 895 (375.9) | 986 (355)

2. Secondary Outcome: Tmax - Time of Occurrence of Cmax
Description: Tmax - time of occurrence of Cmax following an oral single-dose of 50 mg OPC administered alone or 1.5 h after last 1 g Paracetamol administration.
Time Frame: before and ½, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hour post-OPC dose
Measure: Mean (Full Range); unit: hours
Groups:
- Opicapone Alone: Opicapone, OPC, BIA 9-1079
- Opicapone Plus Paracetamol: Opicapone, OPC, BIA 9-1079 Paracetamol, acetominphen
Arm/Group | Opicapone Alone | Opicapone Plus Paracetamol
Number analyzed (Participants) | 28 | 28
hours | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]

3. Secondary Outcome: AUC0-t - Area Under the Plasma Concentration-time Curve (AUC) From Time Zero to the Last Sampling Time at Which the Drug Concentration Was at or Above the Lower Limit of Quantification
Description: AUC0-t - area under the plasma concentration-time curve (AUC) from time zero to the last sampling time following an oral single-dose of 50 mg OPC administered alone or 1.5 h after last 1 g Paracetamol administration
Time Frame: before and ½, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hour post-OPC dose
Measure: Mean (Standard Deviation); unit: ng.h/mL
Groups:
- Opicapone Alone: Opicapone, OPC, BIA 9-1067 50 mg
- Opicapone Plus Paracetamol: Opicapone, OPC, BIA 9-1067 50 mg Paracetamol, acetominophen, 1 g
Arm/Group | Opicapone Alone | Opicapone Plus Paracetamol
Number analyzed (Participants) | 28 | 28
ng.h/mL | 2416 (884.3) | 2818 (1194)

4. Secondary Outcome: AUC0-∞ - Area Under the Plasma Concentration-time Curve (AUC) From Time Zero to Infinity.
Description: AUC0-∞ - AUC from time 0 to infinity following an oral single-dose of 50 mg OPC administered alone or 1.5 h after last 1 g Paracetamol administration.
Time Frame: before and ½, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hour post-OPC dose
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Opicapone Alone | Opicapone Plus Paracetamol
Number analyzed (Participants) | 28 | 28
ng.h/mL | 2451 (882) | 2850 (1188)

ADVERSE EVENTS:
Arm/Group | Opicapone Alone | Opicapone Plus Paracetamol
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 1/28 | 1/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Opicapone Alone (N=28) | Opicapone Plus Paracetamol (N=28)
Nasopharyngitis (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other